CLINICAL TRIAL: NCT01732380
Title: A Multicenter Randomized Phase-II Study Of Raltitrexed/Oxaliplatin Plus Radiotherapy Versus Radiotherapy In Subjects With Inoperable Esophageal Cancer
Brief Title: A Phase-II Study Of Raltitrexed/Oxaliplatin Plus Radiotherapy Versus Radiotherapy In Subjects With Inoperable Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First People's Hospital of Lianyungang (Other)
Collaborators: The East Hospital of Lianyungang (Unknown); Donghai People's Hospital (Other); People's Hospital of Ganyu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1stPeopleLianyungang
Record Dates: First submitted 2012-11-14; First posted 2012-11-22 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Inoperable Esophageal Cancer Stage I-III
MeSH Terms: interventions — raltitrexed; Oxaliplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiotherapy (Active Comparator): Radiotherapy 2.0Gy/day, 5 times/week,6 weeks In Subjects With Inoperable esophageal cancer
  Interventions: Radiation: Radiotherapy
- Raltitrexed/Oxaliplatin Plus Radiotherapy (Experimental): Raltitrexed 2.5mg/㎡ d1,Oxaliplatin 100mg/㎡ d1,q21d Plus Radiotherapy 2.0Gy/day, 5 times/week,6 weeks In Subjects With Inoperable esophageal cancer
  Interventions: Drug: Raltitrexed; Drug: Oxaliplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Raltitrexed
  Other Names: TOMUDEX; Sai Wei Jian
  Arms: Raltitrexed/Oxaliplatin Plus Radiotherapy
Drug: Oxaliplatin
  Other Names: Eloxatin
  Arms: Raltitrexed/Oxaliplatin Plus Radiotherapy
Radiation: Radiotherapy

SUMMARY:
The aim of this study was to compare raltitrexed/oxaliplatin plus radiotherapy versus radiotherapy in subjects with inoperable esophageal cancer.

DETAILED DESCRIPTION:
108 patients were randomized to receive Raltitrexed/Oxaliplatin Plus Radiotherapy (Raltitrexed 2.5mg/㎡ d1,Oxaliplatin 100mg/㎡ d1,q21d Plus Radiotherapy 2.0Gy/day, 5 times/week,6 weeks.)or Radiotherapy ( Radiotherapy 2.0Gy/day, 5 times/week,6 weeks) in subjects with Inoperable esophageal cancer. All patients will receive therapy of six weeks unless disease progression or unacceptable toxicity. Patients were evaluated every 3 months .Progression-Free-Survival was the primary endpoint. Response Rate, Overall survival, toxicity of the therapy are other second endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of inoperable esophageal cancer(squamous cell carcinoma)
* Measurable disease according to RECIST criteria
* Age > 18 years
* WHO performance score < 2
* Estimated life expectancy of > 12 weeks
* Subjects will be considered appropriate to receive systemic chemotherapy and pelvic radiotherapy
* Hematologic function: WBC ≥ 4.0×109/L, PLT ≥ 80×109/L, Hb ≥ 10mg/dL
* Renal function: Cr ≤ 1.25×UNL
* Hepatic function: BIL ≤ 1.5×UNL, ALT/AST ≤ 2.5×UNL
* Documented informed consent to participate in the trial

Exclusion Criteria:

* Subjects with distant metastases
* Pregnancy or breast feeding. Women of childbearing age must use effective contraception
* Serious cardiovascular disease (congestive heart failure, uncontrollable arrhythmia, unstable angina, myocardial infarction, serious heart valve disease, resistant hypertension)
* Evidence of bleeding diathesis or serious infection
* pregnant or lactating woman
* Patient participation in other studies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival | up to 2 years
  Progression-free survival (PFS) is the length of time during and after medication or treatment during which the disease being treated (usually cancer) does not get worse.

SECONDARY OUTCOMES:
Response Rate | up to 2 years
  Response rate (RR) is a figure representing the percentage of patients whose cancer shrinks (termed a partial response, PR) or disappears after treatment (termed a complete response, CR) . In simpler terms RR=PR+CR.

OTHER OUTCOMES:
Overall survival | up to 2 years
  People in a study or treatment group who are still alive for a certain period of time after they were diagnosed with or started treatment for a disease, such as cancer. The overall survival is often stated as a five-year survival, which means people in a study or treatment group who are alive five years after their diagnosis or the start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Jiang, Doctor, Study Chair — The First People's Hospital of Lianyungang
Locations (1):
- The First People's Hospital of Lianyungang, Lianyungang, Jiangsu, China

REFERENCES:
- [Background] Courrech Staal EF, Aleman BM, Boot H, van Velthuysen ML, van Tinteren H, van Sandick JW. Systematic review of the benefits and risks of neoadjuvant chemoradiation for oesophageal cancer. Br J Surg. 2010 Oct;97(10):1482-96. doi: 10.1002/bjs.7175. PMID 20645400
- [Background] Gebski V, Burmeister B, Smithers BM, Foo K, Zalcberg J, Simes J; Australasian Gastro-Intestinal Trials Group. Survival benefits from neoadjuvant chemoradiotherapy or chemotherapy in oesophageal carcinoma: a meta-analysis. Lancet Oncol. 2007 Mar;8(3):226-34. doi: 10.1016/S1470-2045(07)70039-6. PMID 17329193
- [Background] McKenzie S, Mailey B, Artinyan A, Metchikian M, Shibata S, Kernstine K, Kim J. Improved outcomes in the management of esophageal cancer with the addition of surgical resection to chemoradiation therapy. Ann Surg Oncol. 2011 Feb;18(2):551-8. doi: 10.1245/s10434-010-1314-7. Epub 2010 Sep 14. PMID 20839062
- [Background] Seitz JF, Bennouna J, Paillot B, Gamelin E, Francois E, Conroy T, Raoul JL, Becouarn Y, Bertheault-Cvitkovic F, Ychou M, Nasca S, Fandi A, Barthelemy P, Douillard JY. Multicenter non-randomized phase II study of raltitrexed (Tomudex) and oxaliplatin in non-pretreated metastatic colorectal cancer patients. Ann Oncol. 2002 Jul;13(7):1072-9. doi: 10.1093/annonc/mdf183. PMID 12176786
- [Background] Cascinu S, Graziano F, Ferrau F, Catalano V, Massacesi C, Santini D, Silva RR, Barni S, Zaniboni A, Battelli N, Siena S, Giordani P, Mari D, Baldelli AM, Antognoli S, Maisano R, Priolo D, Pessi MA, Tonini G, Rota S, Labianca R. Raltitrexed plus oxaliplatin (TOMOX) as first-line chemotherapy for metastatic colorectal cancer. A phase II study of the Italian Group for the Study of Gastrointestinal Tract Carcinomas (GISCAD). Ann Oncol. 2002 May;13(5):716-20. doi: 10.1093/annonc/mdf091. PMID 12075739